CLINICAL TRIAL: NCT06898801
Title: Neonatal INtubation After "Just-in-time" Audiovisual Training: a Randomised Controlled Trial
Brief Title: An Educational Intervention to Improve the Success of Intubation in Newborns Using a Video Laryngoscope by Reducing the Time the Procedure Takes.
Acronym: NINJA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College Dublin (Other)
Collaborators: National Maternity Hospital, Ireland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: EC44.2024
Record Dates: First submitted 2025-03-06; First posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-02

CONDITIONS: Respiratory Distress Syndrome, Newborn; Endotracheal Intubation; Neonatal Intubation Performance; Prematurity; Neonate; Education, Medical
Keywords: Just-in-Time; Neonatal intubation; Teaching
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn; Premature Birth

STUDY DESIGN:
Intervention Model Description: Shortly before an intubation, a neonate for intubation will be randomised in 1:1 ratio to "Just-in-Time" intervention or none. Randomisation will be stratified by gestational age category: <32 week gestational age (GA) or >32 weeks GA. Allocations will be in sealed opaque envelopes in random order according to gestational age strata. Allocation envelopes will be stored in a dedicated box in the Neonatal Intensive Care Unit (NICU). One randomisation will be carried out for each intubation encounter regardless of number of attempts. Each baby will only be included in the study once. The intubator and team will not be blinded to group assignment as masking will not be possible. Investigators will not be blinded. Outcome assessors will be blinded to the randomisation group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Just-in-Time Intervention (Experimental): The primary intubator, supervising clinician and intubation assistant or nurse will view the brief "Just-in-time" video once, immediately prior to performing the intubation with a video laryngoscope. The decision to intubate an infant and who will perform the intubation will be made by the clinical team. Other aspects of the procedure, for example premedications, use of pre-intubation checklist will not change from standard practice.
  Interventions: Other: Just-in-time video training
- Control (No Intervention): Intubation will be carried out as per current standard practice with supervision of trainee by senior clinician or initial intubation by senior clinician.

INTERVENTIONS:
Other: Just-in-time video training — A "Just-in-time" educational video was designed and produced by the investigating team. Content of the video includes;
  * Environmental set up and patient positioning
  * Equipment preparation including stylet insertion
  * Description of internal anatomy of airway
  * Suggested instructional language for supervisors
  * Example footage of an intubation
  * Tips and common pitfalls
  * Guidance for intubation assistant on how to perform "cricoid" pressure
  Arms: Just-in-Time Intervention

SUMMARY:
This research focuses on one of the most common problems in newborn medicine: breathing difficulties. Breathing problems are the most common reason for admission to our neonatal unit at the National Maternity Hospital. When a baby has serious breathing difficulty, inserting a breathing tube to place them on a ventilator can be lifesaving. A breathing tube must be placed through the vocal cords into the windpipe (trachea). A device called a laryngoscope is placed in a patients mouth to allow the doctor to see the vocal cords and insert the tube correctly.

The skill of placing this breathing tube (intubation) is important for doctors and specialists to learn so that they can confidently perform it in an emergency.

In the past, doctors had more opportunities during their training to learn and practice this with supervision from seniors. In recent years, babies, thankfully, need to be intubated less frequently and doctors working hours are better regulated. As a result, junior doctors have less chances to perform this skill. There is a need to improve how we teach the procedure of intubating babies to doctors in training to meet the needs of trainees today.

The investigators want to perform a study to help teach doctors in training how to perform intubation of a newborn using a video laryngoscope. The team are looking to assess if showing a short educational video to the doctor and team just before performing an intubation using a video laryngoscope will reduce the time the procedure takes. This is called a "Just-in-Time" video. The investigators aim to demonstrate a benefit by performing a randomised control trial. This means that when a baby requires intubation as decided by their treating doctors, the team will be randomly allocated to view a "Just-in-Time" video before performing the intubation or not. The investigators will then compare the two groups to see if there is a difference in the total time the procedure takes.

DETAILED DESCRIPTION:
Performing an urgent intubation on a critically ill newborn can be stressful and daunting. It is a vital, life-saving skill for not only neonatologists but paediatricians who may be faced with the rare scenario of an unwell newborn in respiratory distress. Neonatal intubation remains a mandatory competency of the higher speciality training scheme in General Paediatrics ( Royal College of Physicians of Ireland.) This is in line with paediatric training in the UK and Europe and neonatal intubation competency remains a concern not only in Ireland but worldwide. Teaching neonatal intubation via an apprenticeship model needs to be balanced with the need to minimise risk to babies of prolonged or repeated attempts. Paediatric and neonatal trainees can struggle to achieve competency in this skill as advances in perinatal care such as non-invasive ventilation, less invasive surfactant methods and avoidance of universal intubation for meconium have decreased the number of routine intubations performed. With greater numbers of doctors and advanced neonatal nurse practitioners and fewer working hours, the number of intubation opportunities for trainees continues to fall. Even for more experienced practitioners it can be challenging to maintain intubation competency.

The teaching of skills to paediatricians and neonatologists needs to adapt to the changing nature of training. "Just-in-Time" (JiT) educational interventions have been studied in a variety of simulated and clinical environments to improve training or increase success of uncommonly performed procedures by providing a brief educational intervention shortly before performing the procedure . A study by Gizicki et al applied this concept to neonatal intubation in the clinical setting. They randomised 65 residents performing intubation to receive a Just-in-Time manikin based low fidelity simulation session or a 5-minute video just before performing an intubation. They did not demonstrate a difference in overall intubation success rates between these groups although intubation success rates in both groups were higher than baseline. Intubation in this study was performed using both direct and video laryngoscopy. It has been demonstrated that video laryngoscopy (VL) improves neonatal intubation success, but the method of intubation differs from standard laryngoscopy and there is a learning curve for operators using this device initially. Given that video laryngoscopic intubation is likely to become the standard of care, there is a need to train operators to use this device correctly in order to benefit from its greater utility.

A recent study performed in the National Maternity Hospital by Ni Chathasaigh et al examined video recordings of neonatal intubations using VL. The VAN (Video laryngoscopic Analysis of Neonatal Intubations) study recorded the external environment in addition to the internal VL views of the baby's airway. Analysis of these videos highlights common features of successful and unsuccessful attempts. Using the lessons from the VAN study, the investigators propose a study of a novel "Just-in-Time" educational video to improve intubation performance by reducing the total time required from insertion of the laryngoscope to successful intubation. The "Just-in-Time" video will supplement an intubation checklist and will concentrate on the key aspects of intubation; anatomy, intubator position, cricoid pressure, laryngoscopic technique and supervisor instructions. The "Just-in-Time" video will be directed at the intubator, supervisor and assisting nurse.

ELIGIBILITY:
Inclusion Criteria:

Neonates of any age or gestation who require endotracheal intubation in the Neonatal Intensive Care Unit in the National Maternity Hospital during the study period.

Exclusion Criteria:

* Neonates with an upper airway malformation.
* If it is deemed by the treating clinical team that the clinical scenario does not allow time for the intervention e.g. cardiac arrest

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Total laryngoscopy time in seconds | 24 months
  An intubation attempt is defined as the introduction of the laryngoscope blade into the mouth with the intention of inserting an endotracheal tube (ETT), regardless of whether an ETT was inserted. Laryngoscopy time is the time from insertion of the laryngoscope blade into the mouth during an intubation attempt until removal of the blade, regardless of whether an ETT was successfully inserted. Total laryngoscopy time is defined as the cumulative duration of laryngoscopy time of all intubation attempts undertaken until ETT is inserted and confirmed by exhaled carbon dioxide detection or the procedure is abandoned.

SECONDARY OUTCOMES:
Number of intubation attempts | 24 months
  The number of times the laryngoscope blade is inserted into the mouth with the intention of inserting an endotracheal tube (ETT), regardless of whether an ETT was inserted in one encounter until correct placement of ETT tube, confirmed by exhaled carbon dioxide detection, or procedure abandoned
Duration of each attempt | 24 months
  Duration in seconds of each intubation attempt in an encounter defined as insertion of laryngoscope into the mouth with the intention of inserting an endotracheal tube (ETT), regardless of whether an ETT was inserted.
Lowest heart rate during attempt | 24 months
  Lowest heart rate measured on bedside monitor during intubation attempt (defined above)
Lowest oxygen saturation during attempt | 24 months
  Lowest oxygen saturation measured measured on bedside monitor during intubation attempt (defined above)
Chest compressions during procedure | 24 months
  If chest compressions are required during the intubation
Adrenaline administration during procedure | 24 months
  If bolus adrenaline administration is required during intubation procedure
Oral trauma | 24 months
  If oral trauma is sustained during an intubation
Crossover to alternative operator | 24 months
  Where there are multiple intubation attempts in an encounter, if the practitioner performing intubation is substituted for another for one or more of the attempts

CONTACTS AND LOCATIONS:
Overall Officials: Anna E Curley, Principal Investigator — Department of Neonatology, National Maternity Hospital. University College Dublin; Eoin O'Currain, Principal Investigator — Department of Neonatology, National Maternity Hospital. University College Dublin
Locations (1):
- Department of Neonatology, The National Maternity Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] O'Keeffe AG, Ambler G, Barber JA. Sample size calculations based on a difference in medians for positively skewed outcomes in health care studies. BMC Med Res Methodol. 2017 Dec 2;17(1):157. doi: 10.1186/s12874-017-0426-1. PMID 29197347
- [Background] Kothari R, Hodgson KA, Davis PG, Thio M, Manley BJ, O'Currain E. Time to desaturation in preterm infants undergoing endotracheal intubation. Arch Dis Child Fetal Neonatal Ed. 2021 Nov;106(6):603-607. doi: 10.1136/archdischild-2020-319509. Epub 2021 Apr 30. PMID 33931396
- [Background] Foran J, Moore CM, Ni Chathasaigh CM, Moore S, Purna JR, Curley A. Nasal high-flow therapy to Optimise Stability during Intubation: the NOSI pilot trial. Arch Dis Child Fetal Neonatal Ed. 2023 May;108(3):244-249. doi: 10.1136/archdischild-2022-324649. Epub 2022 Oct 28. PMID 36307187
- [Background] Ni Chathasaigh CM, Dunne EA, Geraghty LE, O'Donnell CPF, O'Currain E, Curley AE. Video analysis of neonatal intubations using video laryngoscopy: a prospective comparison of clinical practice with resuscitation guidelines. Arch Dis Child Fetal Neonatal Ed. 2025 Aug 19;110(5):479-484. doi: 10.1136/archdischild-2024-327723. PMID 39832821
- [Background] O'Shea JE, Loganathan P, Thio M, Kamlin COF, Davis PG. Analysis of unsuccessful intubations in neonates using videolaryngoscopy recordings. Arch Dis Child Fetal Neonatal Ed. 2018 Sep;103(5):F408-F412. doi: 10.1136/archdischild-2017-313628. Epub 2017 Nov 10. PMID 29127153
- [Background] Corder W, Nelin T, Ades AM, Flibotte J, Laverriere E, Daly Guris R, Soorikian L, Foglia EE. Association between video laryngoscopy characteristics and successful neonatal tracheal intubation: a prospective study. Arch Dis Child Fetal Neonatal Ed. 2024 Dec 20;110(1):91-95. doi: 10.1136/archdischild-2024-326992. PMID 38951016
- [Background] Ni Chathasaigh CM, O'Currain E, Curley AE. Variations in newborn airway management. Ir Med J. 2023 May 18;116(5):776. No abstract available. PMID 37555533
- [Background] Lingappan K, Neveln N, Arnold JL, Fernandes CJ, Pammi M. Videolaryngoscopy versus direct laryngoscopy for tracheal intubation in neonates. Cochrane Database Syst Rev. 2023 May 12;5(5):CD009975. doi: 10.1002/14651858.CD009975.pub4. PMID 37171122
- [Background] Riva T, Engelhardt T, Basciani R, Bonfiglio R, Cools E, Fuchs A, Garcia-Marcinkiewicz AG, Greif R, Habre W, Huber M, Petre MA, von Ungern-Sternberg BS, Sommerfield D, Theiler L, Disma N; OPTIMISE Collaboration. Direct versus video laryngoscopy with standard blades for neonatal and infant tracheal intubation with supplemental oxygen: a multicentre, non-inferiority, randomised controlled trial. Lancet Child Adolesc Health. 2023 Feb;7(2):101-111. doi: 10.1016/S2352-4642(22)00313-3. Epub 2022 Nov 24. PMID 36436541
- [Background] Geraghty LE, Dunne EA, Ni Chathasaigh CM, Vellinga A, Adams NC, O'Currain EM, McCarthy LK, O'Donnell CPF. Video versus Direct Laryngoscopy for Urgent Intubation of Newborn Infants. N Engl J Med. 2024 May 30;390(20):1885-1894. doi: 10.1056/NEJMoa2402785. Epub 2024 May 5. PMID 38709215
- [Background] Gizicki E, Assaad MA, Masse E, Belanger S, Olivier F, Moussa A. Just-In-Time Neonatal Endotracheal Intubation Simulation Training: A Randomized Controlled Trial. J Pediatr. 2023 Oct;261:113576. doi: 10.1016/j.jpeds.2023.113576. Epub 2023 Jun 21. PMID 37353151
- [Background] McKay J, Wasserman M, Monuteaux MC, Hirsch AW, Nagler J. Just-in-time procedural training for pediatric emergency medicine trainees: A randomized educational interventional trial. AEM Educ Train. 2023 Jun 22;7(3):e10886. doi: 10.1002/aet2.10886. eCollection 2023 Jun. PMID 37361189
- [Background] Braga MS, Tyler MD, Rhoads JM, Cacchio MP, Auerbach M, Nishisaki A, Larson RJ. Effect of just-in-time simulation training on provider performance and patient outcomes for clinical procedures: a systematic review. BMJ Simul Technol Enhanc Learn. 2015 Oct 5;1(3):94-102. doi: 10.1136/bmjstel-2015-000058. eCollection 2015. PMID 35515199
- [Background] O'Shea JE, Scrivens A, Edwards G, Roehr CC. Safe emergency neonatal airway management: current challenges and potential approaches. Arch Dis Child Fetal Neonatal Ed. 2022 May;107(3):236-241. doi: 10.1136/archdischild-2020-319398. Epub 2021 Apr 21. PMID 33883207